CLINICAL TRIAL: NCT06904560
Title: The Relation Between BSS Solution Temperature and Endothelial Cells and Post Phaco Discomfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Mahmoud,MD, assistant professor of ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: sohag-med-25-1-5PD
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Corneal Diseases
Keywords: cornea, cataract
MeSH Terms: conditions — Corneal Diseases; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Other): patients underwent phacoemulsification , balanced saline solution at room temperature will be used for irrigation
  Interventions: Other: phacoemulsification
- group 2 (Experimental): patients underwent phacoemulsification , balanced saline solution with low (cold ) temperature will be used for irrigation
  Interventions: Other: phacoemulsification

INTERVENTIONS:
Other: phacoemulsification — one group with BSS at room temperature and the other group with cold BSS

SUMMARY:
patients underwent phacoemulsification , balanced saline solution used during the operation will be at room temperature in one group and cool 2.7 c in the other group. the patients will be followed for 3 months after phacoemulsification regarding corneal endothelial cells and anterior segment inflammatory signs

DETAILED DESCRIPTION:
patients underwent phacoemulsification , balanced saline solution used during the operation will be at room temperature in one group and cool 2.7 c in the other group. the patients will be followed for 3 months after phacoemulsification regarding corneal endothelial cells and anterior segment inflammatory signs

ELIGIBILITY:
Inclusion Criteria:

* patients with cataract
* more than 40 years
* no glaucoma
* no retinal abnormalities
* no retinal abnormalities

Exclusion Criteria:

patients with corneal diseases patients less than 40 patients with previous eye surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
endothelial cell count | 3 months

SECONDARY OUTCOMES:
incidence of anterior segment inflammation | 3 months
  incidence of anterior segment inflammation including conjunctival hypremia or corneal edema

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months